CLINICAL TRIAL: NCT03589495
Title: Safety and Efficacy of Adding Intravenous N-acetyl Cysteine to Parenteral L-alanyl L-glutamine in Hospitalized Patients Undergoing Colon Surgeries
Brief Title: Safety and Efficacy of Adding Intravenous N-acetyl Cysteine in Colon Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada Hussein, Principal Investigator, and clinical pharmacist in Ain Shams hospitals, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 79
Record Dates: First submitted 2018-06-15; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- N acetylcysteine group (Active Comparator): N Acetyl L Cysteine IV bolus (100 mg/kg dissolved in dextrose5%) infused over 15 minutes, followed by continuous infusion of 50mg/kg/day dissolved in dextrose 5% starting 1hr before induction of anesthesia, and continued for 48 hours after operation
  Interventions: Drug: N Acetyl L Cysteine
- placebo group (Placebo Comparator): received equal volume of dextrose 5% administrated at the same rate and duration as in the study group as a placebo
  Interventions: Other: dextrose 5%

INTERVENTIONS:
Drug: N Acetyl L Cysteine — 100 mg/kg n acetyl cysteine dissolved in dextrose5%
  Arms: N acetylcysteine group
Other: dextrose 5%
  Arms: placebo group

SUMMARY:
The use of antioxidant agents in the prevention or decreasing the severity of postoperative systemic inflammatory response syndrome after colonic surgeries adopted nowadays. Therefore, it is of interest to investigate safety and efficacy of administrating short term intravenous (IV) N acetyl cysteine as add on to l alany l glutamine and total parenteral nutrition on the marker of oxidative stress malondialdehyde and anti- inflammatory marker tumor necrosis factor alpha in patients undergoing colonic surgeries through a prospective, randomized, double blinded, controlled clinical trial

DETAILED DESCRIPTION:
A prospective, randomized, double blinded, controlled clinical trial will be carried out on 60 patients, who will admit to the critical care unit, Ain Shams hospitals, Cairo, Egypt, following colon surgeries. Before the start of the study, eligible patients were randomized using computer generated list in order to allocate participants to either Group I (n acetyl cysteine group) or Group II (control group) in an equal manner No medication will take before the surgery and only oral fluids were allowed on the day before the operation. All eligible patients underwent bowel preparation with oral 1.745 g/ 30 ml magnesium citrate, and phosphate containing enema on the day before surgery. All patients received the general anesthesia with endotracheal intubation and muscle relaxant.

Data management and analysis were performed using the Statistical Package for Social Sciences (SPSS) software for Windows version 18

ELIGIBILITY:
Inclusion Criteria:

* need for ICU admission after colonic surgery
* requirement of total parenteral nutrition for at least 5 days due to failure of or contraindication for enteral nutrition
* signing a written informed consent.

Exclusion Criteria:

* patients with persistent hemodynamic instability (systolic blood pressure <80 mm Hg), renal impairment, hepatic insufficiency, severe or uncontrolled sepsis, persistent metabolic acidosis, head trauma,and heart failure
* any sensitivity to components of L-alanyl L-glutamine (Dipeptiven®, Fresenius Kabi, Germany) or N acetyl cysteine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07-30 (Actual); Primary Completion 2016-10-15 (Actual); Study Completion 2016-10-15 (Actual)

PRIMARY OUTCOMES:
assessing a change in the level of tumor necrosis factor alpha (TNF alpha) as ant-inflammatory marker reflecting n acetyl cysteine efficacy | Venous blood samples were obtained before surgery (baseline evaluation), and on day two after surgery for measuring changes in TNF ALPHA
  TNF alpha was measured using ELISA technique
assessing a change in the level of malondialdehyde as antioxidant marker in the venous blood sample reflecting n acetyl cysteine efficacy | Venous blood samples were obtained before surgery (baseline evaluation), and on day two after surgery for measuring changes in malondialdehyde level
  malondialdehyde was measured using colorimetric method for assay

SECONDARY OUTCOMES:
measuring safety of N acetyl cysteine (adverse effects) | from the beginning of the study till the patient is discharged from the hospital(up to one week)
  recording any adverse effects that may appear

CONTACTS AND LOCATIONS:
Overall Officials: manal elhammsy, prof, Study Director — Ain Shams University , faculty of pharmacy

IPD SHARING:
Plan to Share IPD: Yes
All the individual participant data will be stored on the computer and will be available on request only
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: it will be available once the trial ends, and for 3 months after publication
Access Criteria: data will be available on request

REFERENCES:
- [Derived] Hamamsy ME, Bondok R, Shaheen S, Eladly GH. Safety and efficacy of adding intravenous N-acetylcysteine to parenteral L-alanyl-L-glutamine in hospitalized patients undergoing surgery of the colon: a randomized controlled trial. Ann Saudi Med. 2019 Jul-Aug;39(4):251-257. doi: 10.5144/0256-4947.2019.251. Epub 2019 Aug 5. PMID 31381364